CLINICAL TRIAL: NCT05437289
Title: A Phase I Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD7442 in Healthy Chinese Adults
Brief Title: A Study to Evaluate the Safety and Tolerability of AZD7442 in Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D8850C00007
Record Dates: First submitted 2022-06-09; First posted 2022-06-29 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Coronavirus Disease 2019 (COVID-19); Healthy Volunteer
Keywords: Coronavirus; COVID-19; AZD7442; Evusheld; LAAB; tixagevimab; AZD8895; cilgavimab; AZD1061
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 300 mg AZD7442 IM (Experimental): Administration of a single dose of 300 mg AZD7442 (150 mg AZD8895 and 150 mg AZD1061) sequentially by intramuscular (IM) injection.
  Interventions: Drug: AZD7442 IM
- 300mg placebo IM (Placebo Comparator): Administration of placebo with dose match to AZD7442 in the same cohort sequentially by intramuscular (IM) injection.
  Interventions: Drug: Placebo IM
- 600 mg AZD7442 IM (Experimental): Administration of a single dose of 600 mg AZD7442 (300 mg AZD8895 and 300 mg AZD1061) sequentially by intramuscular (IM) injection.
  Interventions: Drug: AZD7442 IM
- 600mg placebo IM (Placebo Comparator): Administration of placebo with dose match to AZD7442 in the same cohort sequentially by intramuscular (IM) injection.
  Interventions: Drug: Placebo IM
- 300 mg AZD7442 IV (Experimental): co-administration of a single dose of 300 mg AZD7442 (150 mg AZD8895 and 150 mg AZD1061) by intravenous (IV) infusion.
  Interventions: Drug: AZD7442 IV
- 300mg placebo IV (Placebo Comparator): co-administration of a single dose of placebo in equivalent volume by intravenous (IV) infusion.
  Interventions: Drug: Placebo IV
- 600 mg AZD7442 IV (Experimental): co-administration of a single dose of 600 mg AZD7442 (300 mg AZD8895 and 300 mg AZD1061) by intravenous (IV) infusion.
  Interventions: Drug: AZD7442 IV
- 600mg placebo IV (Placebo Comparator): co-administration of a single dose of placebo in equivalent volume by intravenous (IV) infusion.
  Interventions: Drug: Placebo IV

INTERVENTIONS:
Drug: AZD7442 IM — In cohort 1, participants will be randomized to receive 300 mg AZD7442 (150 mg AZD8895 and 150 mg AZD1061) administered sequentially as direct gluteal IM injections.
  Other Names: AZD7442
  Arms: 300 mg AZD7442 IM
Drug: Placebo IM — In cohort 1, participants will be randomized to receive placebo with dose match to AZD7442 in the same cohort administered sequentially as direct gluteal IM injections.
  Other Names: Placebo
  Arms: 300mg placebo IM
Drug: AZD7442 IM — In cohort 2, participants will be randomized to receive 600 mg AZD7442 (300 mg AZD8895 and 300 mg AZD1061) administered sequentially as direct gluteal IM injections.
  Other Names: AZD7442
  Arms: 600 mg AZD7442 IM
Drug: Placebo IM — In cohort 2, participants will be randomized to receive placebo with dose match to AZD7442 in the same cohort administered sequentially as direct gluteal IM injections.
  Other Names: Placebo
  Arms: 600mg placebo IM
Drug: AZD7442 IV — In cohort 3, participants will be randomized to receive 300 mg AZD7442 (150 mg AZD8895 and 150 mg AZD1061) mixed in IV bag co-administered as a single IV infusion.
  Other Names: AZD7442
  Arms: 300 mg AZD7442 IV
Drug: Placebo IV — In cohort 3, participants will be randomized to receive placebo with dose match to AZD7442 in the same cohort as a single IV infusion.
  Other Names: Placebo
  Arms: 300mg placebo IV
Drug: AZD7442 IV — In cohort 4, participants will be randomized to receive 600 mg AZD7442 (300 mg AZD8895 and 300 mg AZD1061) mixed in IV bag co-administered as a single IV infusion.
  Other Names: Evusheld
  Arms: 600 mg AZD7442 IV
Drug: Placebo IV — In cohort 4, participants will be randomized to receive placebo with dose match to AZD7442 in the same cohort as a single IV infusion.
  Other Names: Placebo
  Arms: 600mg placebo IV

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of AZD7442 in Healthy Chinese Adults. vs. placebo

DETAILED DESCRIPTION:
A Phase I Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD7442 in healthy Chinese participants 18 to 55 years of age, approximately 60 participants will be randomised in a 4:1 ratio to either AZD7442 or placebo, administered by intramuscular (IM) injection or intravenous (IV) infusion, and approximately 479 days in duration for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 55 years of age
2. Healthy by medical history, physical examination, and baseline safety laboratory tests
3. Negative results of both SARS-CoV-2 qRT-PCR and serology tests within 14 days prior to randomisation.
4. Contraceptive within 365 days post dosing

Exclusion Criteria:

1. Medical condition:

   * Known hypersensitivity to monoclonal antibody (mAb) or investigational product (IP) component.
   * Acute illness including fever on the day prior to or day of dosing.
   * Any other significant disease increase the risk to participant study.
2. Laboratory related:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > upper limit of normal (ULN), or alkaline phosphatase (ALP) or TBL (total bilirubin) > 1.5 × ULN
   * Serum creatinine > ULN
   * Haemoglobin < lower limit normal (LLN)
   * Platelet count < LLN
   * White blood cell or neutrophil count outside normal reference ranges
   * Other laboratory significantly abnormal in the screening panel that, in the opinion of the investigator, will increase participants risk or might confound analysis of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From day 1 to approximately 15 months after administration (through Day 451).
  To evaluate the safety and tolerability of AZD7442 administered IM or IV to healthy Chinese participants 18 to 55 years of age.
Incidence of serious adverse events (SAEs) | From day 1 to approximately 15 months after administration (through Day 451).
  To evaluate the safety and tolerability of AZD7442 administered IM or IV to healthy Chinese participants 18 to 55 years of age.
Incidence of adverse event of special interests (AESIs) | From day 1 to approximately 15 months after administration (through Day 451).
  To evaluate the safety and tolerability of AZD7442 administered IM or IV to healthy Chinese participants 18 to 55 years of age.
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of white blood cell (WBC) count, red blood cell (RBC) count.
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of sodium, potassium, urea/blood urea nitrogen (BUN), calcium, phosphate, glucose, c-reactive protein (CRP).
Number of participants with abnormal Coagulation test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of prothrombin time, activated partial thrombin time (aPTT).
Number of participants with abnormal urinalysis | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of glucose, protein, and blood.
Number of participants with abnormal ECG readings | From day 1 to approximately 15 months after administration (through Day 451).
  Results for PR interval, QRS duration, QT interval, QTcF interval, and RR interval will be analyzed.
Number of participants with abnormal vital signs | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of systolic blood pressure (mm Hg), diastolic blood pressure (mm Hg).
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of neutrophils absolute count, lymphocytes absolute count, monocytes absolute count, eosinophils absolute count, Platelets, Reticulocytes absolute count.
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of haemoglobin (Hb).
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of haematocrit (HCT).
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of mean corpuscular volume (MCV).
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of mean corpuscular haemoglobin (MCH).
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transpeptidase (GGT), creatine kinase.
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of creatinine, total bilirubin, conjugated bilirubin.
Number of participants with abnormal laboratory test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of albumin.
Number of participants with abnormal Coagulation test results | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of international normalised ratio (INR).
Number of participants with abnormal ECG readings | From day 1 to approximately 15 months after administration (through Day 451).
  Results for heart rate will be analyzed.
Number of participants with abnormal vital signs | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of pulse rate (beats per minute), respiratory rate (breaths per minute).
Number of participants with abnormal vital signs | From day 1 to approximately 15 months after administration (through Day 451).
  Measurement of body temperature (in degree Celsius).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Research Site, Guangzhou
  - Research Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home